CLINICAL TRIAL: NCT03938545
Title: ASCEND GO-2: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled Study of RVT-1401 for the Treatment of Patients With Active, Moderate to Severe Graves' Ophthalmopathy
Brief Title: ASCEND GO-2: Study of RVT-1401 for the Treatment of Participants With Active, Moderate to Severe Graves' Ophthalmopathy ( GO )
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on premature unblinding of treatment allocations necessitated by program-wide review
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RVT-1401-2001
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Graves' Ophthalmopathy (GO)
Keywords: IMVT-1401; Graves' Orbitopathy; Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen A-RVT-1401 (Experimental): Regimen A= RVT-1401 680 mg weekly for 12 weeks
  Interventions: Drug: RVT-1401 (Administered via subcutaneous injection)
- Regimen B-RVT-1401 (Experimental): Regimen B= RVT-1401 340 mg weekly for 12 weeks
  Interventions: Drug: RVT-1401 (Administered via subcutaneous injection)
- Regimen C-RVT-1401 (Experimental): Regimen C= RVT-1401 255 mg weekly for 12 weeks
  Interventions: Drug: RVT-1401 (Administered via subcutaneous injection)
- Placebo (Placebo Comparator): for 12 weeks
  Interventions: Other: Placebo (Administered via subcutaneous injection)

INTERVENTIONS:
Drug: RVT-1401 (Administered via subcutaneous injection) — RVT-1401 is a fully human anti-neonatal Fc receptor (FcRn) monoclonal antibody.
  Arms: Regimen A-RVT-1401; Regimen B-RVT-1401; Regimen C-RVT-1401
Other: Placebo (Administered via subcutaneous injection) — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the current study is to assess the efficacy and safety/tolerability of three dose regimens of RVT-1401 in the treatment of active, moderate to severe GO participants. In addition, the study is designed to characterize the effect of RVT-1401 exposure on reduction in anti-TSHR IgG

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Clinical diagnosis of Graves' disease with hyperthyroidism associated with active, moderate to severe Graves' Ophthalmopathy (GO) with a Clinical Activity Score (CAS) ≥4 for the most severely affected eye at Screening and Baseline (on the 7-item scale).
3. Onset of active GO within 9 months of screening.
4. Moderate-to-severe active GO (not sight-threatening but has an appreciable impact on daily life), usually associated with one or more of the following: lid retraction ≥2 millimeters (mm), moderate or severe soft tissue involvement, proptosis ≥3 mm above normal for race and gender, and/or inconstant or constant diplopia.
5. Other, more specific inclusion criteria are defined in the protocol

Exclusion Criteria:

1. Use of any steroid (intravenous, oral, steroid eye drops) for the treatment of GO or other conditions within 3 weeks prior to Screening. Steroids cannot be initiated during the trial. Exceptions include topical and inhaled steroids which are allowed.
2. Use of rituximab, tocilizumab, or any monoclonal antibody for immunomodulation within the past 9 months prior to Baseline.
3. Total IgG level <6 grams per liter (g/L) at Screening.
4. Absolute neutrophil count <1500 cells per meter squared (cells/mm^3) at Screening.
5. Participants with decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months at Screening.
6. Previous orbital irradiation or surgery for GO.
7. Other, more specific exclusion criteria are defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (12):
  - Multispecialty Aesthetic Clinical Research Organziation (MACRO), Beverly Hills, California
  - Doheny Eye Center UCLA, Pasadena, California
  - University of Miami Miller School of Medicine Bascom Palmer Eye Institute, Miami, Florida
  - University of Iowa Hospitals & Clinics - Eye Clinic, Iowa City, Iowa
  - University of Michigan - Kellogg Eye Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine - Center for Advanced Medicine (CAM) - Eye Center, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health & Science University (OHSU) - Casey Eye Institute (CEI)-Marquam Hill, Portland, Oregon
  - Eye Wellness Center, Houston, Texas
  - Eyelid Center of Utah, Salt Lake City, Utah
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - Toronto Retina Institute, North York, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Ophthalmology University Center- Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- Germany (3):
  - Universitat Duisburg-Essen, Duisburg
  - Orbitazentrum Frankfurt, Frankfurt am Main
  - Universitätsmedizin Mainz, Mainz
- Italy (3):
  - ARNAS Garibaldi, Presidio di Nesima, Palermo, Catania
  - Fondazione IRCCS Cà Granda-Ospedale Maggiore Policlinico, Milan
  - Unità Operativa di Endocrinologia 2, Azienda Ospedaliero-Universitaria Pisana, Pisa
- Spain (3):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Centro de Oftalmologia Barraquer, Barcelona
  - University Hospital Ramon y Cajal, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 96 participants were screened, of which 65 participants were enrolled and randomized into the study. The total duration of the study was up to 20 weeks.
Groups:
- RVT-1401 680 mg/Week: Participants received a RVT-1401 680 milligram (mg) subcutaneous (SC) injection weekly for 12 weeks.
- RVT-1401 340 mg/Week: Participants received a RVT-1401 340 mg SC injection weekly for 12 weeks.
- RVT-1401 255 mg/Week: Participants received a RVT-1401 255 mg SC injection weekly for 12 weeks.
- Placebo: Participants received a matching placebo SC injection weekly for 12 weeks.
Period: Overall Study
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
Started | 18 | 19 | 10 | 18
Completed | 10 | 14 | 7 | 13
Not Completed | 8 | 5 | 3 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 6 | 4 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 10 | 18 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (9.03) | 52.4 (8.08) | 44.3 (12.61) | 46.1 (12.47) | 47.8 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 8 | 14 | 50
  Male | 3 | 6 | 2 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 17 | 17 | 10 | 18 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 17 | 18 | 10 | 18 | 63
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Mean Proptosis [Mean (Standard Deviation); unit: Millimeters (mm)] | 22.7 (3.10) | 23.0 (3.97) | 22.3 (2.95) | 22.7 (2.70) | 22.72 (3.19)
Mean Clinical Activity Score (CAS) [Mean (Standard Deviation); unit: Units on a scale] — The CAS (7-item scale) measured the acute signs of inflammation like pain, redness, swelling, and impaired function in Graves' Ophthalmology (GO). One point was given for the presence of each of the parameters assessed. The CAS ranged from 0 to 7. Active GO was defined as a CAS of ≥4. Baseline was the last available assessment prior to time of the first dose unless it was specified otherwise and was identified as Day 1. A negative change from baseline represented clinical improvement.
  Units on a scale | 4.8 (0.86) | 5.1 (0.94) | 4.9 (0.99) | 5.2 (1.04) | 5.0 (0.94)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Proptosis Response at Week 13
Description: Proptosis was assessed using an exophthalmometer. A proptosis response was defined as having at least a 2 millimeter (mm) reduction in study eye proptosis without a deterioration (at least a 2 mm increase) in the fellow eye at the same visit. The study eye was defined as the most severely affected eye at the baseline visit.
Time Frame: Baseline; Week 13
Population: Intent-to-Treat (ITT) Population: All randomized participants who received at least one dose of RVT-1401 or placebo and had 1 post-baseline visit. Participants with proptosis assessment at Week 13 were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
Number analyzed (Participants) | 10 | 13 | 6 | 12
Percentage of participants | 30.0 | 30.8 | 0 | 8.3
Statistical Analysis 1: Comparison: RVT-1401 680 mg/Week vs Placebo; Test type: Superiority; p = 0.1993, Cochran-Mantel-Haenszel — p-values were obtained from a Mantel-Haenszel test stratified by smoking status at baseline comparing RVT-1401 680 mg/Week group to placebo; Risk Difference (RD) = 21.4, 95% CI 2-sided [-11.3 to 54.1] — The risk difference was obtained from a weighted average of the difference within each stratum using Cochran Mantel-Haenszel weights
Statistical Analysis 2: Comparison: RVT-1401 340 mg/Week vs Placebo; Test type: Superiority; p = 0.1016, Cochran-Mantel-Haenszel — p-values were obtained from a Mantel-Haenszel test stratified by smoking status at baseline comparing RVT-1401 340 mg/Week group to placebo; Risk Difference (RD) = 24.2, 95% CI 2-sided [-4.8 to 53.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: RVT-1401 255 mg/Week vs Placebo; Test type: Superiority; p = 0.2963, Cochran-Mantel-Haenszel — p-values were obtained from a Mantel-Haenszel test stratified by smoking status at baseline comparing RVT-1401 255 mg/Week group to placebo; Risk Difference (RD) = -8.3, 95% CI 2-sided [-24.0 to 7.3] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (SAEs)
Description: AEs - any untoward medical occurrences in a participant, temporally associated with use of a medicinal product, whether or not considered related to the product. Clinically significant changes determined by the Investigator such as vital signs, ECGs, and clinical laboratory values were also reported as AEs. TEAE is defined as an AE that starts on or after the first dose of the study drug and before 30 days after the last dose of the study drug. SAEs were defined as any untoward medical occurrences that: resulted in death; were life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in disability/incapacity; were congenital anomaly/birth defects; were important medical events that may have jeopardized the participant or may have required medical or surgical intervention; invasive or malignant cancers; and development of drug dependency or drug abuse.
Time Frame: From Baseline up to Week 20
Population: Safety Population: All randomized participants who received at least one dose of either RVT-1401 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
Number analyzed (Participants) | 18 | 19 | 10 | 18
Participants
  TEAEs | 16 | 16 | 8 | 16
  SAEs | 0 | 0 | 1 | 0

3. Secondary Outcome: Least Square Mean Percent Change From Baseline in Binding Anti-thyroid-stimulating Hormone Receptor (TSHR) Antibody Levels to Week 13
Description: Binding Anti-TSHR antibody serum levels are directly associated with GO clinical features. Baseline was the last available assessment prior to the time of the first dose unless it was specified otherwise and was identified as Day 1. A negative change from baseline in binding anti-TSHR antibody levels indicated therapeutic benefit.
Time Frame: Baseline and Week 13
Population: ITT Population. Participants with binding anti-TSHR serum assessments at Week 13 were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
Number analyzed (Participants) | 10 | 13 | 6 | 12
Percent change | -64.605 [-87.006 to -42.205] | -69.663 [-89.272 to -50.054] | -41.843 [-70.070 to -13.616] | -4.520 [-25.580 to 16.539]
Statistical Analysis 1: Comparison: RVT-1401 680 mg/Week vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -60.085, 95% CI 2-sided [-88.857 to -31.313]
Statistical Analysis 2: Comparison: RVT-1401 340 mg/Week vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -65.143, 95% CI 2-sided [-91.927 to -38.358]
Statistical Analysis 3: Comparison: RVT-1401 255 mg/Week vs Placebo; Test type: Superiority; p = 0.0284, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -37.323, 95% CI 2-sided [-70.455 to -4.190]

4. Secondary Outcome: Least Square Mean Percent Change From Baseline in Total IgG Levels
Description: Blood samples we collected to determine total IgG levels. Baseline was the last available assessment prior to the time of the first dose unless it was specified otherwise and was identified as Day 1. A negative change from baseline in the IgG levels indicated therapeutic benefit.
Time Frame: Baseline and Week 13
Population: ITT Population: Participants with evaluable data were included for the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
Number analyzed (Participants) | 10 | 13 | 6 | 12
Percent change | -79.101 [-86.444 to -71.757] | -65.103 [-71.687 to -58.519] | -57.934 [-67.216 to -48.651] | -6.098 [-12.948 to 0.753]
Statistical Analysis 1: Comparison: RVT-1401 680 mg/Week vs Placebo; Week 13; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -73.003, 95% CI 2-sided [-82.309 to -63.697]
Statistical Analysis 2: Comparison: RVT-1401 340 mg/Week vs Placebo; Week 13; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -59.005, 95% CI 2-sided [-67.821 to -50.190]
Statistical Analysis 3: Comparison: RVT-1401 255 mg/Week vs Placebo; Week 13; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -51.836, 95% CI 2-sided [-62.660 to -41.012]

5. Secondary Outcome: Least Square Mean Percent Change From Baseline in IgG Subclasses 1, 2, 3 and 4
Description: Blood samples were collected to determine IgG 1,2,3 and 4 levels. Baseline was the last available assessment prior to the time of the first dose unless it was specified otherwise and was identified as Day 1. A negative change from baseline in the IgG levels indicated therapeutic benefit.
Time Frame: Baseline and Week 13
Population: ITT Population. Participants with evaluable data were included for the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
Number analyzed (Participants) | 9 | 12 | 5 | 9
Percent change
  IgG1 | -82.040 [-90.757 to -73.323] | -68.141 [-75.721 to -60.561] | -67.784 [-79.273 to -56.294] | -0.550 [-9.307 to 8.207]
  IgG2 | -75.346 [-84.395 to -66.297] | -53.678 [-62.077 to -45.280] | -53.879 [-65.648 to -42.110] | -0.481 [-9.392 to 8.431]
  IgG3 | -88.260 [-98.901 to -77.619] | -65.211 [-74.336 to -56.085] | -66.182 [-79.856 to -52.508] | 0.503 [-9.907 to 10.914]
  IgG4 | -68.559 [-77.456 to -59.663] | -55.391 [-63.131 to -47.651] | -52.916 [-64.774 to -41.059] | 0.163 [-9.167 to 9.493]
Statistical Analysis 1: Comparison: RVT-1401 680 mg/Week vs Placebo; IgG1; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -81.490, 95% CI 2-sided [-93.203 to -69.777]
Statistical Analysis 2: Comparison: RVT-1401 340 mg/Week vs Placebo; IgG1; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -67.591, 95% CI 2-sided [-78.562 to -56.620]
Statistical Analysis 3: Comparison: RVT-1401 255 mg/Week vs Placebo; IgG1; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -67.233, 95% CI 2-sided [-81.073 to -53.394]
Statistical Analysis 4: Comparison: RVT-1401 680 mg/Week vs Placebo; IgG2; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -74.865, 95% CI 2-sided [-86.898 to -62.832]
Statistical Analysis 5: Comparison: RVT-1401 340 mg/Week vs Placebo; IgG2; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -53.198, 95% CI 2-sided [-64.799 to -41.596]
Statistical Analysis 6: Comparison: RVT-1401 255 mg/Week vs Placebo; IgG2; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -53.398, 95% CI 2-sided [-67.552 to -39.245]
Statistical Analysis 7: Comparison: RVT-1401 680 mg/Week vs Placebo; IgG3; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -88.764, 95% CI 2-sided [-103.039 to -74.489]
Statistical Analysis 8: Comparison: RVT-1401 340 mg/Week vs Placebo; IgG3; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -65.714, 95% CI 2-sided [-78.742 to -52.686]
Statistical Analysis 9: Comparison: RVT-1401 255 mg/Week vs Placebo; IgG3; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -66.685, 95% CI 2-sided [-83.157 to -50.214]
Statistical Analysis 10: Comparison: RVT-1401 680 mg/Week vs Placebo; IgG4; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -68.722, 95% CI 2-sided [-80.877 to -56.568]
Statistical Analysis 11: Comparison: RVT-1401 340 mg/Week vs Placebo; IgG4; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -55.554, 95% CI 2-sided [-67.182 to -43.926]
Statistical Analysis 12: Comparison: RVT-1401 255 mg/Week vs Placebo; IgG4; Test type: Superiority; p < 0.001, ANCOVA; The model included baseline value of the corresponding parameter, smoking stratum, and treatment group as covariates; Least Square Mean Difference = -53.079, 95% CI 2-sided [-67.948 to -38.210]

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 20
Description: TEAE is defined as an AE that starts on or after the first dose of the study drug and before 30 days after the last dose of the study drug.
Arm/Group | RVT-1401 680 mg/Week | RVT-1401 340 mg/Week | RVT-1401 255 mg/Week | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 1/10 | 0/18
Other Adverse Events (participants affected / at risk) | 16/18 | 16/19 | 8/10 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVT-1401 680 mg/Week (N=18) | RVT-1401 340 mg/Week (N=19) | RVT-1401 255 mg/Week (N=10) | Placebo (N=18)
Optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVT-1401 680 mg/Week (N=18) | RVT-1401 340 mg/Week (N=19) | RVT-1401 255 mg/Week (N=10) | Placebo (N=18)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 9 (9) | 9 (9) | 3 (3) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema migrans (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroxine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroxine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspraxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 5 (5) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to a safety finding (hypercholesterolemia).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03938545/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03938545/SAP_001.pdf